CLINICAL TRIAL: NCT05241392
Title: An Open, Single-arm, Phase 1 Study to Evaluate the Safety/Preliminary Effectiveness and Determine the Maximal Tolerated Dose of B7-H3-targeting CAR-T Cell Therapy in Treating Recurrent Glioblastomas
Brief Title: Safety and Efficacy Study of Anti-B7-H3 CAR-T Cell Therapy for Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yang Zhang, Clinical Professor, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TX103T-IG005
Record Dates: First submitted 2022-01-13; First posted 2022-02-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: a "3+3" design is used to determine Maximum Tolerated Dose (MTD) and the recommended phase 2 dose (RP2D)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T cell therapy (Experimental): Dose-escalation phase:
  A "3+3" dose-escalation design is used to determine MTD & R2PD. Anti-B7-H3 autologous CAR-T cells were given biweekly to patients at the following doses for each cycle, and 4 cycles as one course. Dose1: 3 patients at a dose of 20 million cells for each cycle. Dose 2: 3 patients at a dose of 60 million cells for each cycle. Dose 3: 3 patients at a dose of 150 million cells for each cycle. Dose 4: 3 patients at a dose of 450 million cells for each cycle. Dose 5: 3 patients at a dose of 900 million cells for each cycle.
  R2PD confirmation phase:
  Determine the R2PD based on the results from the previous dose-escalation study; Treat another 12 patients with anti-B7-H3 autologous CAR-T cells biweekly at the R2PD to further confirm the safety of R2PD.
  At each dose phase, if the patients show tolerate and response to the treatment, these patients would receive several courses of treatment at PI's discretion.
  Interventions: Biological: B7-H3-targeting CAR-T cells

INTERVENTIONS:
Biological: B7-H3-targeting CAR-T cells — Patients will be treated with anti-B7-H3 autologous CAR-T cells that are delivered into the intracranial tumor resection cavity or ventricular system using an Ommaya device.

SUMMARY:
This is an open, single-arm, dose-escalation and multiple-dose study to evaluate the safety, tolerability and preliminary effectiveness of B7-H3-targeting Chimeric Antigen Receptor-T (CAR-T) cell therapy on patients with recurrent glioblastomas. The study also plan to explore the Maximum Tolerated Dose (MTD) and determine the Recommended Phase II Dose (RP2D) of the CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-75 years (including 18 and 75 years old)；
2. Patients with relapsed glioblastoma, as confirmed by positron emission tomography (PET) or histologic pathology；
3. A >= 30% staining extent of B7-H3 in his/her primary/recurrent tumor tissue by the immunochemical method;
4. Karnofsky scale score>=50
5. Availability in collecting peripheral blood mononuclear cells (PBMCs) ；
6. Adequate laboratory values and adequate organ function;
7. Patients with childbearing/fathering potential must agree to use highly effective contraception；

Exclusion Criteria:

1. Pregnant or breastfeeding females；
2. Contraindication to bevacizumab；
3. Within 5 days before the CAR-T cell infusion, subjects receiving systemic administration of steroids with dosage more than 10mg/d prednisone or the equivalent doses of other steroids ( not including inhaled corticosteroid)；
4. Comorbid with Other uncontrolled malignancy；
5. Active immunodeficiency virus (HIV) or hepatitis B virus or hepatitis C virus or tuberculosis infection;
6. Subjects receiving the placement of a carmustine slow-release wafer within 6 months before the enrollment;
7. Autoimmune diseases;
8. Receiving long-term immunosuppressive treatment after organ transplantation;
9. Severe or uncontrolled psychiatric diseases or condition that could increase adverse events or interfere the evaluation of outcomes;
10. Not recovered from the toxicities or side effects by previous treatment;
11. Subjects who have participated the other interventional trial within one month before the enrollment, or have received other CAR-T cell therapies or gene-modified cell therapy before enrollment.
12. Subjects with medical conditions that affect signing the written informed consent or complying with the research procedures, the medical conditions including, but not limited to cardio-cerebral vascular diseases, renal dysfunction/failure, pulmonary embolism, coagulation disorders, active systemic infection, uncontrolled infection et. al; or patients who are unwilling or unable to comply with the research procedures; these
13. Subjects with other conditions that would interfere trial participation at the investigator's discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLT) | three months post CAR-T cells infusion
  To evaluate the DLT incidence occurred within three months after B7-H3 CAR-T cells infusion
Safety：Incidence and severity of adverse events | three months post CAR-T cells infusion
  To evaluate the possible adverse events occurred within three months after B7-H3 CAR-T cell infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity

SECONDARY OUTCOMES:
Efficacy：Overall survival rate at 12 months | 12 months post CAR-T cells infusion
  The proportion of subjects who have survived for more than 12 months since the diagnosis of recurrent glioblastoma
Efficacy：objective remission rate | 1, 2, 3, 4, 5, 6 months post CAR-T cells infusion
  The proportion of subjects reaching complete remission / partial remission in optimal remission
pharmacokinetics：Cmax | Samples collected pre-injection, and 1, 2, 3, 5, 7, 9, 11,13 days post the first injection; Samples collected pre-injection, and 2, 7, 13 days post re-injections
  observed maximum plasma concentration (Cmax)
pharmacokinetics：Tmax | Samples collected pre-injection, and 1, 2, 3, 5, 7, 9, 11,13 days post the first injection; Samples collected pre-injection, and 2, 7, 13 days post re-injections
  time to reach maximum plasma concentration (tmax)
pharmacokinetics：AUC | Sample taken pre-injection, and 1, 2, 3, 5, 7, 9, 11,13 days post the first injection; Sample taken pre-injection, and 2,7,13 days post re-injections
  area under the plasma concentration-time curve from time zero to 28 days after dosing (AUC(0-28))

CONTACTS AND LOCATIONS:
Overall Officials: Nan Ji, Dr., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Golubovskaya V. CAR-T Cells Targeting Immune Checkpoint Pathway Players. Front Biosci (Landmark Ed). 2022 Apr 2;27(4):121. doi: 10.31083/j.fbl2704121. PMID 35468680